CLINICAL TRIAL: NCT04676893
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-388 in Healthy Subjects
Brief Title: Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-388 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A99_02BE2002
Record Dates: First submitted 2020-12-18; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference-Test (Experimental)
  Interventions: Drug: D418 Tab.; Drug: CKD-388 Tab.
- Test-Reference (Experimental)
  Interventions: Drug: D418 Tab.; Drug: CKD-388 Tab.

INTERVENTIONS:
Drug: D418 Tab. — 1T
  Other Names: Reference
Drug: CKD-388 Tab. — 1T
  Other Names: Test

SUMMARY:
This study is an open-label, randomized, single dose, crossover study to evaluate the pharmacokinetics, safety and tolerability of CKD-388 in healthy subjects

DETAILED DESCRIPTION:
To healthy subjects of fifty-six (56), following treatments are administered dosing in each period and wash-out period is a minimum of 14 days.

Reference drug: D418 Tab. / Test drug: CKD-388 Tab. Pharmacokinetic blood samples are collected up to 72hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, aged between ≥ 19 and ≤ 45 years old at the time of screening.
2. Weight ≥ 50kg, with calculated body mass index (BMI) of ≥ 18.5 and ≤ 29.9 kg/m2

   * BMI = Weight(kg)/ Height(m)2
3. Individuals who agreed proper contraception during the study and did consent to not donation of sperm 1 month after the last dose of Investigational Product (IP) administration
4. Individuals who voluntary decide to participate and agrees in writing to comply with the precautions after hearing and fully understanding the detailed explanation of this clinical tail

Exclusion Criteria:

1. History or presence of clinically significant and sever active cardiovascular, respiratory, hepatobiliary, renal, hematological, gastrointestinal, endocrine, immune, dermatologic, neurologic, or psychiatric disorder.
2. With symptoms indicating acute illness within 28 days prior to the first Investigational Product (IP) administration.
3. Any medical history that may affect drug absorption, distribution, metabolism and excretion.
4. Individuals who had history of hypersensitivity to follow drugs, derivative drugs or others drugs(aspirin and antibiotics etc.) or had history of drug abuse

   * Thiazolidinedione
   * DPP-4 inhibitor
   * Metformin
5. Any clinically significant chronic medical illness.
6. Any genetic disease including galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
7. Individuals with one of the following laboratory test results in screening

   * AST, ALT > UNL (upper normal limit) x 3
   * Creatinine clearance ≤ 80 mL/min
   * In ECG result, QTc > 450 msec
   * hCG(+) (only women)
8. Individuals who had positive test results at HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL.
9. Use of any prescription drugs within 14 days prior to study drug administration.
10. Use of over-the-counter medications and herbal preparations within 7 days prior to study drug administration.
11. History of any clinically significant allergic reaction (However, mild allergic rhinitis or allergic dermatitis which do not required medication may be allowed).
12. Individuals who cannot eat standard meal provided from clinical trial center.
13. Donation of blood within 60 days prior to study drug administration or apheresis within 20 days prior to the first IP administration.
14. Individuals who had received a blood transfusion within 30 days prior to study drug administration.
15. Exposure to any investigational drug within 6 months prior to the first IP administration.
16. Individuals taking any drugs inducing or inhibiting drug metabolizing enzymes including barbiturates within 30 days prior to the first IP administration.
17. Individuals who had consumed grapefruit juice > 5cups/day or caffeine > 5cups/day within 30 days prior to the first IP administration or who cannot stopping consume grapefruit juice or caffeine during clinical study.
18. Individuals who had drinking (alcohol > 30 g/day) within 30 days prior to the first IP administration or who cannot stop drinking.
19. Heavy smoking (more than 10 cigarettes/day) within 30 days prior to screening or who cannot quit smoking during clinical study.
20. Pregnant or women who may be pregnant
21. Subjects having been deemed inappropriate for the trial as determined by the investigator.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-02-26 (Estimated); Primary Completion 2021-05-11 (Estimated); Study Completion 2021-05-18 (Estimated)

PRIMARY OUTCOMES:
AUCt of CKD-388, D418 | Pre-dose (0 hour), post-dose 0.17, 0.33, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72 hours
  Area under the CKD-388/D418 concentration in blood-time curve from zero to final
Cmax of CKD-388, D418 | Pre-dose (0 hour), post-dose 0.17, 0.33, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72 hours
  The maximum CKD-388/D418 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No